CLINICAL TRIAL: NCT02038257
Title: Prospective Open Label Parallel Study Comparing Use of Carbon Dioxide Laser Versus Dermabrasion for Denuding Epithelium and Collagen Dressing Versus Vaseline Impregnated Gauze for the Melanocyte Keratinocyte Transplant Procedure
Brief Title: Comparative Study Using Dermabrasion vs CO2 Laser & Collagen Dressing vs Vaseline Gauze in MKTP
Acronym: MKTP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Iltefat Hamzavi, Principle Investigator, Henry Ford Health System
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8082
Record Dates: First submitted 2014-01-10; First posted 2014-01-16 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Vitiligo; Depigmented Scars; Depigmentation
MeSH Terms: conditions — Vitiligo | interventions — Lasers, Gas; Dermabrasion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- MKTP with CO2 Laser/Collagen Dressing (Active Comparator): Each Subject will have a depigmented patch of skin treated with MKTP using the carbon dioxide laser for de-epithelialization and a collagen dressing for the wound dressing.
  Interventions: Procedure: MKTP (melanocyte keratinocyte transplant procedure); Device: Collagen Dressing; Device: Carbon Dioxide Laser
- MKTP with CO2 laser/vaseline gauze (Active Comparator): Each subject will have a depigmented patch of skin treated with MKTP using the carbon dioxide laser for de-epithelialization and vaseline impregnated gauze as the wound dressing.
  Interventions: Procedure: MKTP (melanocyte keratinocyte transplant procedure); Device: Vaseline Impregnated Gauze; Device: Carbon Dioxide Laser
- MKTP with dermabrasion/collagen dressing (Active Comparator): Each subject will have a depigmented patch of skin treated with MKTP using dermabrasion for de-epithelialization and a collagen dressing for the wound dressing.
  Interventions: Procedure: MKTP (melanocyte keratinocyte transplant procedure); Device: Collagen Dressing; Device: Dermabrasion
- MKTP with dermabrasion/vaseline gauze (Active Comparator): Each subject will have a depigmented patch of skin treated with MKTP using dermabrasion for de-epithelialization and vaseline impregnated gauze as a wound dressing.
  Interventions: Procedure: MKTP (melanocyte keratinocyte transplant procedure); Device: Vaseline Impregnated Gauze; Device: Dermabrasion

INTERVENTIONS:
Procedure: MKTP (melanocyte keratinocyte transplant procedure) — Each subject will have the melanocyte keratinocyte transplant procedure on 4 distinct areas using the two different techniques being studied (carbon dioxide laser and dermabrasion) and the two different dressings being studied (vaseline impregnated gauze and collagen dressing).
  Other Names: MKTP
Device: Collagen Dressing — Each subject will have MKTP on 4 distinct areas. Two of these areas will be dressed with a collagen dressing.
  Arms: MKTP with CO2 Laser/Collagen Dressing; MKTP with dermabrasion/collagen dressing
Device: Vaseline Impregnated Gauze — Each subject will have MKTP on 4 distinct areas of depigmented skin. Two of these areas will be dressed with vaseline impregnated gauze.
  Arms: MKTP with CO2 laser/vaseline gauze; MKTP with dermabrasion/vaseline gauze
Device: Carbon Dioxide Laser — Each subject will have MKTP on 4 distinct areas of depigmented skin. Two of these areas will be de-epithelialized using a carbon dioxide laser.
  Other Names: CO2 laser
  Arms: MKTP with CO2 Laser/Collagen Dressing; MKTP with CO2 laser/vaseline gauze
Device: Dermabrasion — Each subject will have MKTP on 4 distinct areas of depigmented skin. Two of these areas will be de-epithelialized using dermabrasion.
  Arms: MKTP with dermabrasion/collagen dressing; MKTP with dermabrasion/vaseline gauze

SUMMARY:
The purpose of this study is to:

1. Compare two different techniques in the melanocyte keratinocyte transplant procedure: Use of carbon dioxide laser versus use of dermabrasion
2. Compare two different dressings in the melanocyte keratinocyte transplant procedure: vaseline impregnated gauze versus collagen dressing

DETAILED DESCRIPTION:
The melanocyte keratinocyte transplant procedure (MKTP) has been shown to be effective in treating vitiligo and other conditions with depigmented skin. MKTP involves the transplantation of melanocytes and keratinocytes from normal skin onto the depigmented skin in order to repigment the skin.

Both dermabrasion and carbon dioxide lasers have been used effectively in MKTP to denude the epithelium. This study will compare the efficacy of these two techniques.

The study will also compare the efficacy of two different dressings used in MKTP, vaseline impregnated gauze and collagen dressings.

ELIGIBILITY:
Inclusion Criteria:

* Depigmented patches of skin

Exclusion Criteria:

* History of Acral Vitiligo
* Unstable Vitiligo, defined as new areas of depigmentation or enlarging areas of depigmentation within the last 6 months
* History of hypertrophic scarring or keloids
* History of koebnerization (new patches of vitiligo at sites of injury or trauma)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-01; Primary Completion 2018-12 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Vitiligo Assessment Scoring Index (VASI) | 6 months
  Assessment of the percentage of repigmentation and color match of the repigmentation.

SECONDARY OUTCOMES:
Time to De-Epithelialization | Assessed at Visit 1 (Day of Procedure)
  Amount of time needed to de-epithelialize the skin using carbon dioxide laser versus dermabrasion
Pain Severity Scale | Assessed on Visit 1 (Day of Procedure)
  Assess pain experienced on a severity scale from 0-10 during de-epithelialization with carbon dioxide laser versus dermabrasion, and during dressing application with vaseline impregnated gauze versus collagen dressing.

CONTACTS AND LOCATIONS:
Overall Officials: Iltefat H Hamzavi, MD, Principal Investigator — Henry Ford Dermatology
Locations (1):
- Henry Ford Dermatology, Detroit, Michigan, United States